CLINICAL TRIAL: NCT00325390
Title: Double-Blind Parallel Comparison Study of SR25990C Versus Standard Therapy in Japan(Ticlopidine) in Patients With Acute Coronary Syndrome Without ST-Segment Elevation Who Are Planned for Percutaneous Coronary Intervention
Brief Title: Efficacy and Safety in Patients With Acute Coronary Syndrome Without ST-Segment Elevation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Daiichi Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC6720
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Platelet Aggregation Inhibitors; NSTEACS
Keywords: SR25990C; Platelet Aggregation Inhibitors; NSTEACS
MeSH Terms: interventions — Clopidogrel

INTERVENTIONS:
Drug: clopidogrel (SR25990C)

SUMMARY:
To evaluate the efficasy and safety of SR25990C(loading dose:300mg, maintenance dose:75mg/day) in comparison with the standard Japanese treatment(ticlopidine) in patients with acute coronary syndrome without ST-segment elevation and planned for percutaneous coronary intervention(including stenting).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 20, admitted to hospitals with symptoms suspected to represent an acute coronary syndrome defined as unstable angina or acute MI without ST segment elevation greater than 1 mm are eligible for the study if they meet the following criteria:

  * (1)Clinical history consistent with new onset or worsening pattern of characteristic ischemic chest pain occurring at rest or with minimal exercise (lasting longer than 5 minutes or requiring sublingual nitroglycerin for the relief of pain within 24 hours before registration).
  * (2)Patients who meet either of following criteria

    * ECG changes compatible with new ischemia [e.g. ST depression (at least 1 mm), T wave inversion (at least 2 mm), or hyperacute peaked T waves in 2 contiguous leads].
    * already elevated CK at least twice the upper limit of normal or CK-MB or Troponin I or T above the upper limit of normal or positive qualitative test for Troponin T.
  * (3)A percutaneous coronary intervention is planned within 96 hours after the first study drug administration

Exclusion Criteria:

* A)Factors that affect participation in study:

  * (1)Previous disabling stroke
  * (2)Previous intracranial hemorrhage or hemorrhagic stroke
  * (3)Severe co-morbid condition such that the patient is not expected to survive 1 month
  * (4)NYHA Class IV heart failure
  * (5)Uncontrolled hypertension
  * (6)Requirement for use of oral anticoagulants, non study antiplatelet agents (including ticlopidine) or NSAIDs (excluding unum sumatur), during study period,
* B)Factors related to ASA and/or ticlopidine treatment:

  * (1)Use of ticlopidine within 1 week prior to randomization
  * (2)History of ASA or ticlopidine intolerance or allergy
  * (3)Contraindications to ASA or ticlopidine

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2004-07

PRIMARY OUTCOMES:
Incidence of effficacy and safety events

SECONDARY OUTCOMES:
Incidence of efficacy or safety events, adverse events, adverse drug reactions and bleeding events・

CONTACTS AND LOCATIONS:
Overall Officials: Yuko HARADA, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan